CLINICAL TRIAL: NCT07357077
Title: The Relationship Between Upper Extremity Anthropometric Measurements and Reaction Time
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, MSc, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: 2024/14-22
Record Dates: First submitted 2026-01-07; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy Persons
Keywords: reaction time; anthropometric measurement; upper extremity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aimed to examine the relationship between upper extremity anthropometric measurements and reaction time in healthy individuals. Also, we aimed to investigate whether there are differences between dominant and non-dominant upper extremity anthropometric measurements and reaction time.

DETAILED DESCRIPTION:
Reaction time is the time between the presentation of a stimulus and the generation of a response. It consists of various processes including sensory processing, information processing, decision-making, and motor response. Reaction time is also affected by various factors such as task complexity, attention level, and the individual's condition. Muscle strength has been shown to affect reaction time in different age groups. Studies in the literature have determined that reaction time is a factor affecting performance in athletes, individuals with orthopedic diseases, and the elderly. Therefore, identifying the factors affecting reaction time is important. We aimed to investigate the relationship between upper extremity anthropometric measurements and reaction time in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-30 years old
* Not having undergone any surgery on the upper or lower extremities

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Having undergone surgery on their upper and lower extremities, Using orthotics Having deformities and contractures Having neurological diseases
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Anthropometric Measurements | Baseline
  Upper extremity length measurements were performed twice and the average score was recorded. Total upper extremity, arm and forearm length measurements were taken with a Harpenden anthropometer. Hand, palmar (palm), thumb, index finger, middle finger, ring finger, little finger, hand width and hand opening length measurements were taken with a digital caliper (Dasqua, Italy).

SECONDARY OUTCOMES:
Reaction time measurement | Baseline
  Reaction time was assessed using the Blazepod device (Blazepod 1.0). A four-LED evaluation panel was used for measurement. Individuals were asked to turn off the LEDs as quickly as possible while in a seated position. The average time between the LEDs turning on and the individuals touching and turning them off the illuminated sensors was recorded by the device in milliseconds for each hand separately. A one-minute rest period was given between tests. The test was conducted twice, and the best score was recorded. The dominant and non-dominant upper extremities were evaluated, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Hüseyin GÜNGÖR, Undergraduate Student, Principal Investigator — Kütahya Health Sciences University; Yusuf ÖZTÜRK, Undergraduate Student, Principal Investigator — Kütahya Health Sciences University; Lütfiye AKKURT, PhD, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)